CLINICAL TRIAL: NCT06728787
Title: Efficacy of Robot-assisted Walking Treatment on Gait Biomechanics, Functional Outcomes, and Quality of Life in Subjects With Hereditary Spastic Paraplegia (HSP)
Brief Title: Robot-assisted Walking Treatment in Hereditary Spastic Paraplegia (HSP)
Status: Recruiting | Type: Observational
Sponsor: IRCCS Eugenio Medea (Other)
Responsible Party: Sponsor
Other Study IDs: GIP 1065
Record Dates: First submitted 2023-10-17; First posted 2024-12-11 (Actual); Last update posted 2025-05-04 (Actual); Status verified 2025-04

CONDITIONS: Hereditary Spastic Paraplegia
MeSH Terms: conditions — Spastic Paraplegia, Hereditary

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Hereditary Spastic Paraplegia (HSP): Patients undergo a combined rehabilitation treatment consisting of 15 sessions on Lokomat and 15 sessions of physical therapy over three weeks for a total of 30 sessions. The same subjects undergo clinical-functional evaluations before, at the end of treatment and after a 3-month follow-up.
  Interventions: Device: Robot-Assisted Gait Training

INTERVENTIONS:
Device: Robot-Assisted Gait Training — 15 sessions of robot-assisted gait training(LOKOMAT)+ 15 session of usual treatment for a total of 30 sessions in three weeks. 45 minutes for each session.

SUMMARY:
Patients will undergo a combined rehabilitation treatment consisting of 15 sessions on Lokomat and 15 sessions of physical therapy over three weeks for a total of 30 sessions. Two sessions/day for 5 days a week. The same subjects will conduct clinical-functional assessments before, at the end of treatment, and after a 3-month follow-up:

3D Gait Analysis with defined protocol (BTSBioenginner); Spastic Paraplegia Rating Scale (SPRS); Six-Minute Walk Test (6MWT), Ten Meters Walk Test (10MWT), Gross Motor Function Measure-88 (GMFM-88) and Berg Balance Scale (BBS); Quality of life questionnaires: Medical Outcome Survey Short Form (SF-36) and ad hoc questionnaire for subjective assessment of symptoms during walking (HSP-SNAP).

This study is part of normal clinical practice and does not involve any changes to the current rehabilitation course for patients.

DETAILED DESCRIPTION:
In the field of rare neurological diseases, familiar spastic paraplegia represents a movement disorder with no specific therapy that can treat the disease or stop its evolution. Therefore, "therapy" is mainly symptomatic, going to act not on the cause of the disorder but on its clinical manifestation. In this context, the definition of effective rehabilitative treatment protocols is extremely important to ensure a qualitatively consistent intake with the goal of containing the functional decline related to the natural history of pathology. The crucial aspect of the disease is represented by alterations in gait pattern resulting in reduced functional skills and negative impact on the subject's quality of life.

Over the past 20 years, robotic technological gait rehabilitation has entered and spread in addition to conventional rehabilitation because of its ability to be highly motivating and engaging, showing itself effective as a complementary therapy. Among the various systems on the market, Lokomat (HOCOMA) is one of the most popular and widely used for treatment in both pediatric and adult populations. The literature is full with works in which Lokomat is used in subjects with neurological disorders (Stroke, Spinal Cord Injury, Infantile Cerebral Palsy) with good results especially in the functional domain. The objective of our study is to evaluate the efficacyof an intensive rehabilitation protocol with Lokomat combined with traditional treatment in a mixed population (pediatric and adult) of subjects with hereditary spastic paraplegia. In addition, follow-up evaluation will allow consideration of the maintenance of the results obtained from the intensive course.

Patients undergo a combined rehabilitation treatment consisting of 15 sessions on Lokomat and 15 sessions of physical therapy over three weeks for a total of 30 sessions. The same subjects undergo clinical-functional evaluations before, at the end of treatment and after a 3-month follow-up:

3D Gait Analysis with defined protocol (BTSBioenginner); Spastic Paraplegia Rating Scale (SPRS); Six-Minute Walk Test (6MWT), Ten Meters Walk Test (10MWT), Gross Motor Function Measure-88 (GMFM-88) and Berg Balance Scale (BBS); Quality of life questionnaires: Medical Outcome Survey Short Form (SF-36) and ad hoc questionnaire for subjective assessment of symptoms during walking (HSP-SNAP).

The proposed study is both retrospective and prospective: 29 subjects have already been included in the retrospective database, and it is hypothesized to collect data from an additional 21 subjects.

The treatment will be able to take place in both inpatient and MAC settings, and the protocol includes performance evaluation through clinical and instrumental assessments in the population of subjects with HSP treated with the Lokomat device at the IRCCS Medea site in Bosisio Parini.

ELIGIBILITY:
Inclusion Criteria:

* genetic or clinical diagnosis of HSP.
* age greater than 4 years and less than 70
* femur length > 23 cm
* ability to walk independently indoors, with or without walking aids.

Exclusion Criteria:

* botulinum toxin injection or lower limb surgery in the previous 6 months
* severe lower limb muscle retractions
* severe osteoporosis
* unhealed skin lesions in lower limbs
* cardiovascular instability
* acute or progressive neurological disorders
* behavioral problemS

Ages: 4 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients affected by a hereditary spasti paraplegia with or without a genetic diagnosis.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2012-01-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Six-Minute Walk Test (6MWT) | T0(pre-training)
  Endurance Test
Six-Minute Walk Test (6MWT) | T1(after 3 weeks of training)
  Endurance Test
Six-Minute Walk Test (6MWT) | T2(3 months after T1)
  Endurance Test

SECONDARY OUTCOMES:
Medical Outcome Survey Short Form (SF-36) | T0(pre-training)
  Questionnaire Quality of Life. 2 index: physical health and mental health. Higher score better health perception.
Hereditary Spastic Paraplegia Self-Notion and Perception (HSP-SNAP) | T0(pre-training)
  Questionnaire Self-Notion and Perception. Scoring: 0-48. Higher score better health.
Spastic Paraplegia Rating Scale (SPRS) | T0(pre-training)
  Severity of the HSP. Score: 0-52. Higher score more severity.
Medical Outcome Survey Short Form (SF-36) | T1(after 3 weeks of training)
  Questionnaire Quality of Life. 2 index: physical health and mental health. Higher score better health perception.
Hereditary Spastic Paraplegia Self-Notion and Perception (HSP-SNAP) | T1(after 3 weeks of training)
  Questionnaire Self-Notion and Perception. Scoring: 0-48. Higher score better health.
Spastic Paraplegia Rating Scale (SPRS) | T1(after 3 weeks of training)
  Severity of the HSP. Score: 0-52. Higher score more severity
Medical Outcome Survey Short Form (SF-36) | T2(3 months after T1)
  Questionnaire Quality of Life. 2 index: physical health and mental health. Higher score better health perception.
Hereditary Spastic Paraplegia Self-Notion and Perception (HSP-SNAP) | T2(3 months after T1)
  Questionnaire Self-Notion and Perception. Scoring: 0-48. Higher score better health.
Spastic Paraplegia Rating Scale (SPRS) | T2(3 months after T1)
  Severity of the HSP. Score: 0-52. Higher score more severity

OTHER OUTCOMES:
3D GAIT ANALYSIS | T0(pre-training),T1(after 3 weeks of training),T2(3 months after T1)
  Analysis of the gait pattern
Ten Meters Walk Test (10MWT) | T0(pre-training),T1(after 3 weeks of training),T2(3 months after T1)
  Gait Velocity Test
Gross Motor Function Measure-88 (GMFM-88) | T0(pre-training),T1(after 3 weeks of training),T2(3 months after T1)
  Pediatric Gross Motor Evaluation. Score:0-264. Higher score more function.
Berg Balance Scale (BBS) | T0(pre-training),T1(after 3 weeks of training),T2(3 months after T1)
  Balance Test. Score:0-56. Higher score better balance.
3D GAIT ANALYSIS | T1(after 3 weeks of training)
  Analysis of the gait pattern
Ten Meters Walk Test (10MWT) | T1(after 3 weeks of training)
  Gait Velocity Test
Gross Motor Function Measure-88 (GMFM-88) | T1(after 3 weeks of training)
  Pediatric Gross Motor Evaluation. Score:0-264. Higher score more function.
Berg Balance Scale (BBS) | T1(after 3 weeks of training)
  Balance Test. Score:0-56. Higher score better balance.
3D GAIT ANALYSIS | T2(3 months after T1)
  Analysis of the gait pattern
Ten Meters Walk Test (10MWT) | T2(3 months after T1)
  Gait Velocity Test
Gross Motor Function Measure-88 (GMFM-88) | T2(3 months after T1)
  Pediatric Gross Motor Evaluation. Score:0-264. Higher score more function.
Berg Balance Scale (BBS) | T2(3 months after T1)
  Balance Test. Score:0-56. Higher score better balance.

CONTACTS AND LOCATIONS:
Locations (1):
- Irccs Eugenio Medea, Bosisio Parini, Italy/lecco, Italy

IPD SHARING:
Plan to Share IPD: No